CLINICAL TRIAL: NCT02946606
Title: A Randomized, Active-controlled, Multiple-dose, Open-label Study to Evaluate the Safety, Tolerability, and Efficacy of the Long-acting Antibody-fused Recombinant Human Growth Hormone (GX-H9) in Adult Growth Hormone Deficiency (AGHD)
Brief Title: A Clinical Study in AGHD to Assess Safety, Tolerability and Efficacy of GX-H9
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX-H9-002
Record Dates: First submitted 2015-08-28; First posted 2016-10-27 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — GX-H9; Human Growth Hormone

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: GX-H9 + Genotropin (Experimental): GX-H9 (weekly dose), Genotropin (daily)
  Interventions: Drug: GX-H9; Drug: Genotropin
- Group 2: GX-H9 + Genotropin (Experimental): GX-H9 (weekly dose), Genotropin (daily)
  Interventions: Drug: GX-H9; Drug: Genotropin
- Group 3: GX-H9 + Genotropin (Experimental): GX-H9 (weekly dose), Genotropin (daily)
  Interventions: Drug: GX-H9; Drug: Genotropin

INTERVENTIONS:
Drug: GX-H9 — Human growth hormone
Drug: Genotropin — Human growth hormone

SUMMARY:
This is a randomized, active-controlled, open-label, sequential dose group, Phase 1b/2 study designed to assess the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of weekly and every other week doses of GX-H9 in the treatment of AGHD.

DETAILED DESCRIPTION:
The subjects who are adequately eligible to attend this clinical trial via screening will be sequentially assigned starting with Group 1. Each group will be comprised of subjects who will receive both GX-H9 and Genotropin, and subjects will be randomly assigned to either GX-H9 and Genotropin in the ratio of 4:1. The treatment will proceed as the proposed group order (Group 1, Group 2, Group 3), and safety and insulin-like growth factor (IGF-1) will be reviewed six weeks after each treatment by the safety monitoring committees before proceeding to the next group.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Is a male or female aged ≥20 and 65 years with AGHD, either adult onset GHD due to hypothalamic pituitary disease or childhood onset GHD that is either idiopathic or due to hypothalamic pituitary disease or due to genetic causes.
2. Has documented confirmation (medical history) of GH deficiency during adulthood by 1 or more growth hormone (GH) stimulation tests, as follows:

   * Insulin tolerance test (peak hGH≤3.0 ng/mL)
   * Arginine + growth-hormone-releasing hormone (peak hGH≤4.0 ng/mL)
3. Has been treated with stable hormonal replacement therapies for deficiencies of other hypothalamo pituitary axes and must have been on an optimized and stable treatment regimen for at least 3 months before screening (free thyroxine [T4] level within normal range at screening). Temporary adjustment of glucocorticoid replacement therapy, as appropriate, is acceptable.
4. Has a screening IGF-1 level of at least 1 standard deviation (SD) score (IGF-1 SD score <1) below the mean IGF-1 level standardized for age and gender according to the central laboratory reference values.
5. Has a BMI of ≥18.0 and 35.0 kg/m2 (both male and female subjects).
6. Has a confirmed negative test result for anti-recombinant human growth hormone (anti-rhGH) antibodies at screening.
7. Must agree to use appropriate contraceptive methods (ie, condoms, cervical cap in conjunction with spermicide, sterilization, and intra uterine device) during the study and for 6 months after the last dose of study drug.
8. Female subjects must have a negative serum pregnancy test result at screening.
9. Must be willing and able to provide written informed consent before performing any study procedures.

Exclusion Criteria:

A subject meeting any of the following criteria will be excluded from the study:

1. Has evidence of growth of pituitary adenoma or other intracranial tumor within the last 12 months which has to be confirmed by computed tomography or magnetic resonance imaging scan (with contrast) within 3 months before screening. (Subjects with inactive remnant intracranial tumors are eligible).
2. Is currently receiving antitumor therapy and has a history of malignancy other than i) cranial tumor or leukemia causing GHD, or ii) fully treated basal cell carcinoma or evidence of active malignancy.
3. Has any clinically significant electrocardiogram (ECG) abnormality at screening.
4. Has evidence of intracranial hypertension at screening.
5. Has uncontrolled diabetes mellitus with diet and exercise, as determined based on glycated hemoglobin (HbA1c) levels ≥7.0% at screening.
6. Has impaired liver function defined as elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.0 × upper limit of normal (ULN).
7. Has impaired kidney function defined as increased serum creatinine levels greater than 1.5 × ULN.
8. Has had active acromegaly within 18 months before screening.
9. Has active carpal tunnel syndrome.
10. Has Prader-Willi syndrome.
11. Has had active Cushing syndrome within 12 months before screening.
12. Has any other major medical conditions, including eg, clinically manifested hypertension, tuberculosis, major surgery within the 3 months before screening, or significantly abnormal laboratory test results (eg, disturbed calcium homeostasis); or any other conditions (eg, acute infections) that may influence drug absorption, metabolism, or excretion, or that may interfere with any study variables in the judgment of the investigator.
13. Has been treated with systemic corticosteroids other than replacement therapy within 3 months before screening.
14. Is a female subject of childbearing potential who is pregnant, breastfeeding, or intends to become pregnant.
15. Has been treated with anabolic steroids other than gonadal steroid replacement therapy within 2 months before screening. Oral estrogen replacement and hormonal contraceptives are not allowed in female subjects. For replacement purposes, transdermal estrogens are permitted in female subjects.
16. Has a history of noncompliance with medications, uncooperativeness, or alcohol/drug abuse.
17. Has a positive result from serology examination for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
18. Has a known or suspected hypersensitivity to rhGH.
19. Has donated blood or had any major blood loss greater than 500 mL within 90 days before screening.
20. Has a history of any medical or psychiatric condition that in the opinion of the investigator would pose a risk for participation in this study or interfere with the compliance needed for this study.
21. Has received an investigational drug or product or has participated in a drug study within 60 days before screening.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
The change in insulin-like growth factor-1 (IGF-1) levels in relation to time and dose strength | 12 weeks

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of GX-H9 in the treatment of AGHD: Area under the curve, AUC0-t | 12 weeks
PK profile of GX-H9 in the treatment of AGHD: Area under the curve, AUC0-inf | 12 weeks
PK profile of GX-H9 in the treatment of AGHD: Area under the curve, AUC0-tau | 12 weeks
PK profile of GX-H9 in the treatment of AGHD: Maximum serum concentration, Cmax | 12 weeks
PK profile of GX-H9 in the treatment of AGHD: The time taken to reach the maximum concentration, Tmax | 12 weeks
PK profile of GX-H9 in the treatment of AGHD: Half-life, t1/2 | 12 weeks
Pharmacodynamic (PD) profile of GX-H9 in the treatment of AGHD: Maximum serum concentration of IGF-1, Cmax | 12 weeks
PD profile of GX-H9 in the treatment of AGHD: Area under curve of IGF-1, AUC0-t | 12 weeks
PD profile of GX-H9 in the treatment of AGHD: Maximum serum concentration of IGFBP-3, Cmax | 12 weeks
PD profile of GX-H9 in the treatment of AGHD: Area under curve of IGFBP-3, AUC0-t | 12 weeks
Data in Physical examination, Vital signs, Electrocardiography, Clinical Laboratory Test Results Related to Investigational Product | 12 weeks
Immunogenicity Test After subcutaneous injection of GX-H9 | 12 weeks
The changes of glucose metabolism indices | 12 weeks
Data in hormonal status of thyroid, estradiol(female), testosterone(male), and cortisol levels | 12 weeks
The lipid parameters as actual values and percent change from baseline (CFB)at week 12: total cholesterol | change from baseline at 12weeks
The lipid parameters as actual values and percent change from baseline (CFB) at week 12: High-density lipoprotein cholesterol | change from baseline at 12weeks
The lipid parameters as actual values and percent change from baseline (CFB) at week 12: low-density lipoprotein cholesterol | change from baseline at 12weeks
The lipid parameters as actual values and percent change from baseline (CFB) at week 12: Triglycerides | change from baseline at 12weeks
The lipid parameters as actual values and percent change from baseline (CFB) at week 12: lipoprotein[a] | change from baseline at 12weeks
The waist circumference as actual values and CFB at week 12 | change from baseline at 12weeks
The hip circumference as actual values and CFB at week 12 | change from baseline at 12weeks
The waist-to-hip ratio as actual values and CFB at week 12 | change from baseline at 12weeks
The BMI as actual values and CFB at week 12 | change from baseline at 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eun Jig Lee, MD, PhD, Principal Investigator — Yonsei University
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No